CLINICAL TRIAL: NCT02481661
Title: A Phase III Randomized Trial of Anatomical Segmentectomy Versus Lobectomy by Minimal Incision for Stage IA Peripheral Non-Small Cell Lung Cancer (≤ 2cm)
Brief Title: Comparison of Lobectomy and Segmentectomy for cT1aN0M0 Peripheral NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- segmentectomy (Experimental): Patients undergo anatomic segmentectomy by minimal incision thoracotomy or thoracoscopy/VATS.
  Interventions: Procedure: segmentectomy
- lobectomy (Active Comparator): Patients undergo lobectomy by minimal incision thoracotomy or thoracoscopy/VATS.
  Interventions: Procedure: segmentectomy

INTERVENTIONS:
Procedure: segmentectomy — segmentectomy in Arm I and lobectomy in Arm II

SUMMARY:
Anatomic segmentectomy may be a less invasive type of surgery than lobectomy for cT1aN0M0 peripheral NSCLC and may retain more pulmonary function. It is not yet known whether anatomic segmentectomy is non-inferior to lobectomy in treating stage IA non-small cell lung cancer. The aim of this study is to investigate whether the outcome of anatomic segmentectomy is similar to lobectomy for peripheral stage IA (≤ 2cm)non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Objective: To compare the outcomes(including 5 year relapse free survival rate, 5 year overall survival rate, retaining pulmonary function and the rates of loco-regional and systemic recurrence ) of patients with peripheral stage IA (≤ 2 cm) non-small cell lung cancer undergoing anatomic segmentectomy vs lobectomy. And to evaluate whether the anatomic segmentectomy is an optimal type of surgery for the patients with peripheral stage IA (≤ 2cm) non-small cell lung cancer (NSCLC).

Outline: This is a multicenter, prospective, randomized open phase III study of anatomic segmentectomy vs lobectomy for the patients with peripheral stage IA (≤ 2cm) non-small cell lung cancer (NSCLC). According to completely random block design, the patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo anatomic segmentectomy by minimal incision thoracotomy or thoracoscopy/VATS.
* Arm II: Patients undergo lobectomy by minimal incision thoracotomy or thoracoscopy/VATS.

Patients will be followed up every 3 months for the first year and then every 6 months for the subsequent 2 years and annually for 5 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70y
2. Preoperative criteria:

   ⅰ)Center of tumor is located in the outer third of the lung field, and the maximal diameter ≤ 2 cm(including coronal, traverse and sagittal view) confirmed by 1mm thin layer contrast-enhanced CT scan.

   ⅱ)no hilar and mediastinal lymph node metastasis verified by mediastinoscope/EBUS.
3. Intraoperative criteria:

   ⅰ)Adenocarcinama or squamous cell carcinoma of lung confirmed by frozen section.

   ⅱ)Lobectomy, single segmentectomy or combined segmentectomy is feasible.

   ⅲ)Confirmation of N0 status by frozen section examination of nodal levels 10 and 13 for segmentectomy, and 10 for lobectomy.
4. ECOG performance status 0-2.
5. No other malignancy within the past 3 years( except for well prognostic malignancy such as basal cell carcinoma of skin, superficial bladder cancer, or carcinoma in situ of the cervix).
6. No prior ipsilateral thoracotomy (prior diagnostic thoracoscopy is allowed).
7. No prior chemotherapy or radiation therapy.
8. Lobectomy is tolerated.
9. Sufficient organ functions.
10. Written informed consent.

Exclusion Criteria:

1. Active bacterial or fungous infection.
2. Simultaneous or metachronous (within the past 5 years) multiple cancers.
3. Interstitial pneumonitis, pulmonary fibrosis, or severe pulmonary emphysema, and can not tolerate lobectomy.
4. Psychosis.
5. Uncontrollable diabetes mellitus.
6. History of severe heart disease.
7. The maximal diameter of GGO≤5mm.
8. N1, N2, or M1a is confirmed postoperatively.
9. Postoperative adjuvant therapy (chemotherapy ,radiotherapy or targeted therapy).
10. Other types of lung cancer such as small cell lung cancer, large cell lung cancer, etc.
11. Confirmation of benign disease by postoperative pathologic examination.
12. Lesion located in the middle lobe.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2015-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | 5 years
  To evaluate the 5 year relapse-free survival (RFS) rate of two groups.

SECONDARY OUTCOMES:
overall survival | 5 years
  To evaluate the 5 year overall survival (OS) rate of two groups.
Pulmonary function | 6 months and 12 months
  to evaluate the pulmonary function as measured by expiratory flow rate of the two groups 6 months and 12 months postoperatively.
the duration of postoperative hospital stay | an expected average of 5 days
  to evaluate the postoperative inpatient days of the two groups.
performance status | 12 months
  to evaluate the postoperative performance status of the two groups by ECOG score standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China